CLINICAL TRIAL: NCT06437600
Title: Immediate Angioplasty For Acute Ischemic Stroke With Severe Intracranial Atherosclerotic Stenosis (MAGIC): A Multicenter, Prospective, Open-label, Blinded Endpoint, Randomized Controlled Trial
Brief Title: Immediate Angioplasty For Acute Ischemic Stroke With Severe Intracranial Atherosclerotic Stenosis
Acronym: MAGIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2024-337-02
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Stroke, Acute Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): Participants will receive immediate angioplasty (with or without stenting) for the culprit vessel and the target residual stenosis should be less than 50%. All participants will receive the best medical treatment (BMT).
  Interventions: Procedure: Immediate angioplasty
- The control group (No Intervention): Participants will receive BMT alone.

INTERVENTIONS:
Procedure: Immediate angioplasty — See arm/group descriptions.
  Arms: The intervention group

SUMMARY:
A multicenter, prospective, open-label, blinded endpoint, randomized controlled trial that aims to evaluate the effect of immediate angioplasty (with or without stenting) for acute ischemic stroke (AIS) with severe intracranial atherosclerotic stenosis (ICAS) in improving the 90-day functional outcome.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, open-label, blinded endpoint, randomized controlled trial designed to evaluate the effect of immediate angioplasty (with or without stenting) for AIS with severe ICAS. The primary outcome is the proportion of patients with a 90-day modified Rankin scale (mRS) of 0-2.

Study intervention: (1) Participants in the intervention group will undergo immediate angioplasty (with or without stenting), and will receive the best medical treatment (BMT) after the procedure. (2) Participants in the control group will receive BMT alone.

This study is anticipated to enroll 412 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Diagnosed with AIS and baseline NIHSS ≥6.
3. Pre-stroke mRS ≤2.
4. Time from symptom onset to randomization ≤ 24 hours; the onset time refers to "Last Known Well" (LKW).
5. Non-contrast CT ASPECTS score ≥6.
6. CTA confirmed severe ICAS (70-99%) of the intracranial segment of the internal carotid artery, or M1 or M2 segment of the middle cerebral artery, and is presumed to be responsible for the stroke.
7. Informed consent signed by the patient or authorized representative.

Exclusion Criteria:

1. Normal diameter of the culprit vessel <2.0 mm.
2. Isolated perforator artery infarction (except for combined cortical hypoperfusion).
3. Hemorrhagic stroke within the past 90 days.
4. Cerebrovascular conditions such as vasculitis, moya-moya disease, arterial inflammatory stenosis, vasospasm, traumatic dissection, etc..
5. Severe calcification at the stenosis site, where expected residual stenosis ≤50% cannot be achieved with procedure.
6. Known cardiac thrombus source (e.g., atrial fibrillation, patent foramen ovale, infective endocarditis).
7. INR >1.7 when using warfarin; coagulation dysfunction or uncorrectable bleeding factors.
8. Platelet count <50×10^9/L.
9. Intracranial hemorrhage confirmed by CT or MRI.
10. Women who are pregnant or breastfeeding.
11. Participation in other intervention clinical trials.
12. Known severe renal insufficiency with glomerular filtration rate <30 ml/min or blood creatinine >220 μmol/L (2.5 mg/dl).
13. Severe allergy to contrast (non-mild rash allergy) or absolute contraindication to iodine contrast.
14. Aortic dissection.
15. Concomitant intracranial tumor (except for meningioma <10mm) or arteriovenous malformation.
16. Severe vascular tortuosity, difficult access for intervention, or inability to complete endovascular treatment.
17. Any active bleeding or recent bleeding in the last 1 month.
18. SBP>185 mmHg or DBP>110 mmHg refractory to treatment.
19. Anticipated life expectancy <3 months (e.g., malignancy, severe cardiopulmonary disease, etc.).
20. Any condition that, in the judgment of the investigator, makes the patient unsuitable for this study or where this study may impose a significant risk to the patient (e.g., inability to understand and/or comply with study procedures and/or follow-up due to psychiatric disorders, cognitive or emotional impairment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The modified Rankin Scale (mRS) 0-2 | 90(±7) days
  The proportion of the mRS 0-2 at 90 days.

SECONDARY OUTCOMES:
The mRS 0-1 | 90(±7) days
  The proportion of the mRS of 0-1 at 90 days.
The mRS 0-3 | 90(±7) days
  The proportion of the mRS of 0-3 at 90 days.
The shift analysis of the mRS distribution | 90(±7) days
  The distribution of the mRS at 90 days.
The change of National Institute of Health Stroke Scale (NIHSS) | 7(±1) days or discharge, whichever came first
  The change of NIHSS from baseline to 7 days or discharge (whichever comes first).
Any new stroke (ischemic/hemorrhagic) or all-cause mortality | within 30 days
  Any new stroke (ischemic/hemorrhagic) or all-cause mortality within 30 days
Any recurrent stroke in the territory of the target artery | within 90 days
  Any recurrent stroke in the territory of the target artery within 90 days
The quality of life | 90(±7) days
  The value of quality of life (EQ-5D-5L) at 90 days.

OTHER OUTCOMES:
SAFETY OUTCOME: Symptomatic intracranial hemorrhage | 24 (±12) hours
  Symptomatic intracranial hemorrhage within 36 hours (according to Heidelberg criteria).
SAFETY OUTCOME: Mortality | 90(±7) days
  Mortality at 90 days.
SAFETY OUTCOME: Any intracranial hemorrhage | 24 (±12) hours
  Any intracranial hemorrhage within 36 hours (according to Heidelberg criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, M.D., Ph.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Yajie Liu, M.D., Ph.D., Principal Investigator — Shenzhen Hospital of Southern Medical University
Locations (2):
- China (2):
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available from Principal Investigators (Prof. Yamei Tang and Prof. Yajie Liu) upon reasonable request 6 months after the trial completion.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the trial completion.
Access Criteria: The IPD will be available from Principal Investigators (Prof. Yamei Tang and Prof. Yajie Liu) upon reasonable request.